CLINICAL TRIAL: NCT03309696
Title: Regulating Homeostatic Plasticity and the Physiological Response to rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 206326
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This prospective, experimental design includes a block randomized, blinded, sham controlled, mixed effects model with sequential assignment to treatment arms (1 or 10 Hz rTMS) and random assignment to the tDCS conditions within each arm. The order of the three experimental conditions within each arm is randomized.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- tDCS and 1 Hz rTMS delivered over TC (Experimental): Participants receive sham and active 2mA tDCS over the temporal cortex (TC) prior to receiving sham and active 1 Hz rTMS (900 rTMS pulses at 110% motor threshold) delivered to the TC. .
  Interventions: Device: sham tDCS and sham rTMS; Device: sham tDCS and active rTMS; Device: active tDCS and active rTMS
- tDCS and 10Hz rTMS delivered over TC (Experimental): Participants receive sham and active 2mA tDCS over the temporal cortex (TC) prior to receiving sham and active 10 Hz rTMS (900 rTMS pulses at 110% motor threshold) delivered to the TC.
  Interventions: Device: sham tDCS and sham rTMS; Device: sham tDCS and active rTMS; Device: active tDCS and active rTMS
- tDCS over DLFC and 1 Hz rTMS over TC (Experimental): Participants receive sham and active 2mA tDCS over the dorsolateral frontal cortex (DLFC) prior to receiving sham and active 1 Hz rTMS (900 rTMS pulses at 110% motor threshold) delivered to the TC.
  Interventions: Device: sham tDCS and sham rTMS; Device: sham tDCS and active rTMS; Device: active tDCS and active rTMS
- tDCS over DLFC and 10 Hz rTMS over TC (Experimental): Participants receive sham and active 2mA tDCS over the dorsolateral frontal cortex (DLFC) prior to receiving sham and active 10 Hz rTMS (900 rTMS pulses at 110% motor threshold) delivered to the TC.
  Interventions: Device: sham tDCS and sham rTMS; Device: sham tDCS and active rTMS; Device: active tDCS and active rTMS

INTERVENTIONS:
Device: sham tDCS and sham rTMS — Both combinations of tDCS and rTMS in this intervention are sham.
  Other Names: transcranial direct current stimulation (tDCS), repetative transcranial magnetic stimulation (rTMS)
Device: sham tDCS and active rTMS — tDCS in this intervention is sham and rTMS is active
  Other Names: transcranial direct current stimulation (tDCS), repetative transcranial magnetic stimulation (rTMS)
Device: active tDCS and active rTMS — Both combinations of tDCS and rTMS in this intervention are active
  Other Names: transcranial direct current stimulation (tDCS), repetative transcranial magnetic stimulation (rTMS)

SUMMARY:
This device-study includes a pilot, physiological investigation of normal human subjects. The aim is to determine how existing non-invasive neuromodulation devices affect brain circuitry as measured by EEG recording. Currently, the application of non-invasive neuromodulation is rarely guided by detailed knowledge of how neural activity is altered in the brain circuits that are targeted for intervention. This gap in knowledge is problematic for interpreting response variability, which is common. To address this gap, the current proposal aims to combine two forms of neuromodulation sequentially, transcranial direct current stimulation (tDCS) and repetitive transcranial magnetic stimulation (rTMS), to regulate homeostatic plasticity prior to rTMS delivery at different frequencies of rTMS. Homeostatic plasticity, the initial activation state of a targeted circuit, is a key determinant of whether rTMS induces long term potentiation (LTP) or long term depression (LTD) Yet, homeostatic plasticity is rarely measured or controlled in rTMS studies. We aim to control homeostatic plasticity by preconditioning the targeted circuits with tDCS prior to rTMS delivery. The protocol included an exploratory aim to examine physiological changes in patients with tinnitus but this aim was not part of the pilot physiological investigation and it could not be completed due to funding limitations.

DETAILED DESCRIPTION:
Background and Rationale: The current proposal aims to combine two forms of neuromodulation, transcranial direct current stimulation (tDCS) and repetitive transcranial magnetic stimulation (rTMS), to regulate homeostatic plasticity prior to rTMS delivery at two different frequencies (1Hz and 10Hz). Homeostatic plasticity, the initial activation state of a targeted circuit, is a theoretical determinant of whether rTMS induces long term potentiation (LTP) or long term depression (LTD).Yet, homeostatic plasticity is rarely measured or controlled in rTMS studies. In a physiological investigation of health subjects, we aim to control homeostatic plasticity by preconditioning the targeted circuits with tDCS prior to rTMS delivery. The justification for this study is that controlling homeostatic plasticity can reduce subject variability and the knowledge gained can be used to optimize rTMS delivery. What is needed to move the field forward is a method for combining tDCS and rTMS and for measuring neuronal responses directly which we aim to establish in this study. The pilot study project will examine the targeted effects of neuromodulation in normal subjects. The brain regions targeted for intervention include auditory areas in the temporal cortex (TC) that process sounds and functionally connected regions of the dorsolateral frontal cortex (DLFC) that mediate sensory habituation. Due to funding limitations, only the 1 Hz rTMS condition could be initiated.

ELIGIBILITY:
Inclusion Criteria:

* complete the informed consent process
* men and women, age: 21-65 years
* negative pregnancy test (female subjects of childbearing age must take a pregnancy test).

Exclusion Criteria:

* a personal or family history of epilepsy,
* severe head injury, aneurysm, stroke, previous cranial neurosurgery,
* sever or recurrent migraine headaches,
* metal implants in the head or neck, a pacemaker,
* pregnancy,
* medications that lower seizure threshold,

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mennemeier, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS and 1 Hz rTMS Delivered Over TC | tDCS Over DLFC and 1 Hz rTMS Over TC | tDCS and 10Hz rTMS Delivered Over TC | tDCS Over DLFC and 10 Hz rTMS Over TC
Started | 5 (All five subjects in this arm were randomize to all sham and active tDCS and rTMS interventions.) | 5 (All five subjects in this arm were randomize to all sham and active tDCS and rTMS interventions.) | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 5 | 0 | 0
Not completed — Analysis of TEP data could not be completed | 0 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the two arms to which subjects were assigned.
Groups:
- tDCS and 1 Hz rTMS Delivered Over TC: Baseline characteristics for participants assigned to the arm that received tDCS and 1Hz rTMS over the temporal cortex.
- tDCS and 1 Hz rTMS Delivered Over DLPF: Baseline characteristics for participants assigned to the arm that received tDCS and 1Hz rTMS over the dorsolateral frontal cortex.
- Total: Total of all reporting groups
Arm/Group | tDCS and 1 Hz rTMS Delivered Over TC | tDCS and 1 Hz rTMS Delivered Over DLPF | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (16.8) | 32 (15.14) | 33.9 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Mean baseline P100 amplitude of the GMFA [Mean (Standard Deviation); unit: µV] — The mean of the P100 amplitude during a baseline recording, before any of the tDCS or rTMS interventions have been introduced. Population: Outcome measures are not reported for the DLPF arm because, due to insufficient resources and the required personnel needed to perform the data cleaning and pipeline analysis, no P100 amplitude data can be reported.
  µV
    number analyzed (Participants) | 5 | 0 | 5
    (all) | 1.29 (0.47) |  | 1.29 (0.47)

OUTCOME MEASURES:

1. Primary Outcome: Log Transformed P100 Amplitude of TEPs From the Global Mean Field Analysis.
Description: TEPs refer to TMS-evoked EEG potentials. The P100 amplitude of TEPs is one means of assessing cortical excitability. The P100 amplitude has been shown to be a reliable metric in studies of healthy subjects. The P100 amplitude is used in this study to assess the excitation state of two regions of interest (ROIs), one in the TC and one in the DLPFC, at each period of TEP recording (i.e., Baseline, Post tDCS, Post rTMS, and 20 minute delay).
Time Frame: Up to 8 weeks
Population: The analyses population is 5 subjects who were assigned to the arm "tDCS and 1 Hz rTMS over the temporal cortex". The group titles reflect sequences of sham and active tDCS and rTMS conditions used to create contrasts for data analysis. Outcome measures are not reported for the DLPF arm because, due to insufficient resources and the required personnel needed to perform the extensive data cleaning and pipeline analysis, no P100 amplitude data can be reported.
Measure: Mean (Standard Deviation); unit: log µV
Groups:
- Sham tDCS Preconditioning: TEPs recorded post sham tDCS but before rTMS.
- Active tDCS Preconditioning: TEPs recorded after active tDCS preconditioning but before rTMS.
- Sham tDCS Preconditioning of Sham rTMS: TEPs recorded after sham tDCS preconditioning and sham rTMS.
- Sham tDCS Preconditioning of Active rTMS: TEPs recorded after sham tDCS preconditioning and active rTMS.
- Active tDCS Preconditioning of Active rTMS: TEPs recorded after active tDCS preconditioning and active rTMS.
Arm/Group | Sham tDCS Preconditioning | Active tDCS Preconditioning | Sham tDCS Preconditioning of Sham rTMS | Sham tDCS Preconditioning of Active rTMS | Active tDCS Preconditioning of Active rTMS
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
log µV | 1.85 (0.71) | 1.26 (0.33) | 1.59 (0.82) | 1.30 (0.58) | 1.11 (0.48)
Statistical Analysis 1: Comparison: Sham tDCS Preconditioning vs Active tDCS Preconditioning; Examines the effect of tDCS preconditioning on P100 amplitudes. The effect size for this comparison was .33 (Cohen's); Test type: Equivalence — A p value of <.0.05 is taken as evidence of nonequivalence; p = .055, Mixed Models Analysis — The p value is not adjusted because it was a planned contrast; Mean Difference (Net) = -.59 — Active tDCS - sham tDCS
Statistical Analysis 2: Comparison: Sham tDCS Preconditioning vs Sham tDCS Preconditioning of Active rTMS; Examines the effect of rTMS on the P100 amplitude. The calculated effect size is .35 (Cohen's); Test type: Equivalence — A p value of <.05 is taken as evidence of nonequivalence; p = 0.0418, Mixed Models Analysis — This p value is not adjusted for multiple comparisons because it was a planned contrast; Mean Difference (Net) = .36 — Sham tDCS - Sham tDCS and Active rTMS
Statistical Analysis 3: Comparison: Sham tDCS Preconditioning of Active rTMS vs Active tDCS Preconditioning of Active rTMS; Examines the additive effect of tDCS preconditioning on the P100 amplitude after rTMS. The effect size for this comparison was 0.14; Test type: Equivalence — A p value less than 0.05 is taken as evidence of nonequivalence; p = 0.40, Mixed Models Analysis — The p value is not adjusted as this was a planned contrast; Mean Difference (Net) = -0.19 — Effect of tDCS preconditioning on active rTMS: active tDCS preconditioning of active rTMS - sham tDCS preconditioning of active rTMS
Statistical Analysis 4: Comparison: Sham tDCS Preconditioning of Sham rTMS vs Active tDCS Preconditioning of Active rTMS; Examines the combined effect of tDCS and rTMS on the P100 amplitude. The effect size for this comparison was .29 (Cohen's); Test type: Equivalence — A p value less than 0.05 is taken as evidence of nonequivalence; p = .086, Mixed Models Analysis — The p value was not adjusted for this planned contrast; Mean Difference (Net) = -0.48 — Active tDCS and Active rTMS - Sham tDCS and Sham rTMS

ADVERSE EVENTS:
Time Frame: Three lab visits over 6 weeks.
Groups:
- Cumulative Report of Adverse Events: Adverse events data were collected irrespective of Arm/Group assignment. Adverse events were coded as either serious/nonserious, expected/unexpected, and related or unrelated to the intervention. There was only 1 adverse event (a mild headache, which was nonserious, expected and related to active rTMS).
Arm/Group | Cumulative Report of Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cumulative Report of Adverse Events (N=10)
Headache (Skin and subcutaneous tissue disorders) | 1 (1) — Mild headache reported after TMS stimulation.

LIMITATIONS AND CAVEATS:
Our pilot study funding ended. Subjects could not be recruited for the 10 Hz rTMS arm. A proposed study of tinnitus patients could not be initiated. Data analysis could only be completed for one arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT03309696/Prot_SAP_000.pdf